CLINICAL TRIAL: NCT02635841
Title: The Compassionate Use of Deferiprone in Patients With Pantothenate Kinase-Associated Neurodegeneration
Brief Title: Compassionate Use of Deferiprone in Patients With PKAN
Status: No longer available | Type: Expanded Access
Sponsor: Chiesi Canada Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: TIRCON2012V1-COMP
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pantothenate Kinase-Associated Neurodegeneration
Keywords: Pantothenate Kinase-Associated Neurodegeneration; PKAN; Neurodegeneration with Brain Iron Accumulation; NBIA; Deferiprone; Ferriprox
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration | interventions — Deferiprone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Deferiprone — Ferriprox (deferiprone) 100 mg/mL oral solution
  Other Names: Ferriprox

SUMMARY:
Patients with pantothenate kinase-associated neurodegeneration (PKAN) who have completed the ApoPharma-sponsored study TIRCON2012V1-EXT and who wish to continue to take deferiprone will be offered the opportunity to receive it on a compassionate basis. Patients will be followed locally by their own neurologist or other appropriate specialist.

DETAILED DESCRIPTION:
Patients with PKAN who have completed both the randomized, blinded, placebo-controlled trial TIRCON2012V1 and its follow-up, the single-arm open-label extension study TIRCON2012V1-EXT, may enroll in this compassionate-use/expanded access program in order to continue receiving the iron chelator deferiprone. Participants in this program will be followed locally by their own neurologist or other appropriate specialist. Patients will take deferiprone oral solution 80 mg/mL at the same dose they were prescribed in the TIRCON2012V1-EXT clinical trial. Safety monitoring of the patients will be performed. At a minimum, the program will continue until the analysis of the currently blinded TIRCON2012V1 trial is completed (approximately Q4 2016), at which time it will be re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Completed study TIRCON2012V1-EXT
2. Able to adhere to program appointments and evaluation schedules
3. Females of childbearing potential must have a negative pregnancy test result at the start of the program, unless the treating physician determines there is no reasonable risk of pregnancy because of significant incapacity. If applicable, they must meet at least one of the following criteria: Use an effective method of contraception during the program and for 30 days following the last dose of deferiprone, OR participate in a non-heterosexual lifestyle, OR have a male sexual partner who has been sterilized, OR be abstinent during the program and for at least 30 days after its completion.
4. Fertile sexually active heterosexual males must agree to use an effective method of contraception during the program and for at least 30 days after its completion
5. Patients and/or their authorized legal representatives must provide signed and dated written informed consent, and minors must additionally sign an assent form as per local regulatory requirements.

Exclusion Criteria:

Patients will be excluded from taking part in the compassionate use program if the treating physician determines the presence of any medical, psychological, or psychiatric condition which in his/her opinion would cause participation in the program to be unwise

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult